CLINICAL TRIAL: NCT06333301
Title: Translational Initiative to Map Epigenetics in Sleep
Acronym: TIME-ZZZ
Status: Not yet recruiting | Type: Observational
Sponsor: Elysium Health (Industry)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: TIME-ZZZ
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Biological Aging
Keywords: Sleep; Chronotype
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TIME-ZZZ: Group will complete several surveys
  Interventions: Other: Surveys

INTERVENTIONS:
Other: Surveys — Group will complete several surveys

SUMMARY:
The primary aim of TIME-ZZZ is to explore the relationship between chronotype, incidence of depression and biological age, and whether individuals working "out-of-phase" with their chronotype are more likely to exhibit signs of depression and accelerated biological aging.

DETAILED DESCRIPTION:
Understanding the relationship between chronotype, depression, and biological age is important in the field of sleep research and mental health. Sleep patterns and their alignment with an individual's internal body clock, or chronotype, have been increasingly recognized as influential factors in various aspects of well-being, including mental health and overall physiological aging. By conducting a study that investigates the potential correlation between chronotype, incidence of depression, and biological age, along with the impact of working "out-of-phase" with one's chronotype, the investigators can shed light on crucial aspects of sleep, mental health, and their interplay with biological aging.

ELIGIBILITY:
Inclusion Criteria:

* Has taken an INDEX test within the last 3 months
* Has registered at least 1 INDEX kit via the Elysium Health website
* Able and willing to provide digital consent to the RSCF, and the TIME-ZZZ Research Subject Consent Form

Exclusion Criteria:

* Consent to participate not given

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2034-04 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Effect of being "out of phase" with chronotype on biological age | At baseline
  Determine whether individuals working "out-of-phase" with their chronotype (from TIME-ZZZ survey responses) exhibit higher rates of biological aging compared to those working within their chronotype

SECONDARY OUTCOMES:
Effect of Chronotype Alignment and Depression Risk in Relation to Rate of Aging | At baseline
  Determine the effect of chronotype alignment and depression risk (from TIME-ZZZ surveys) on biological rate of aging
Identification of DNA methylation markers associated with chronotype | At baseline
  Identify specific DNA methylation markers associated with chronotype (from TIME-ZZZ surveys) thereby providing potential insights into the epigenetic regulation of sleep-wake patterns
Identification of DNA methylation markers associated with depression | At baseline
  Identify specific DNA methylation markers associated with depression (from TIME-ZZZ surveys) potentially shedding light on the underlying epigenetic mechanisms involved in the development and progression of depressive disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Dayle Sampson, PhD, Principal Investigator — Elysium Health; Russell Foster, PhD, Principal Investigator — University of Oxford

IPD SHARING:
Plan to Share IPD: No